CLINICAL TRIAL: NCT01225861
Title: Prospective Study on the Use of Transdermal Analgesic Buprenorphine Patches for Chronic Pain in the UK
Status: Completed | Type: Observational
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 241437
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is the descriptive analysis of incidence & severity of side effects & reasons for discontinuation of the treatment of chronic pain with transdermal analgesic Buprenorphine patches.

DETAILED DESCRIPTION:
750 patients that are treated with transdermal Buprenorphine patches for chronic pain will be included in the study. About 20% of patients are aimed to be patch-naive, ie have received their first prescription of transdermal analgesic patches within 1 month before inclusion in this observational study. Furthermore the study should not include more than 25% of cancer patients that are treated for chronic pain in order to ensure an appropriate mix of patient population.

ELIGIBILITY:
Inclusion Criteria

* Patient age > 18
* Patient is treated with transdermal Buprenorphine
* The patient is able to answer the patient's survey & has an estimated overall survival of minimum 6 months
* The patient gives his/her informed, written consent to participate in the study

Exclusion Criteria

* Patient Age < 18
* Patient has less than 6 months survival expectancy
* Patient is unable to answer the patient survey for whatever reason in any feasible form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing pain. They may be from primary or secondary care.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of side effects | patients observed for 6 months
  Descriptive analysis of incidence and severity of side effects and reasons for discontinuation with Buprenorphine patches. Safety Issue - No

SECONDARY OUTCOMES:
Treatment patterns | patients observed for 6 months
  Insight into patient profiles treatment patterns and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Infirmary, Terrent Institute, Glasgow, United Kingdom

REFERENCES:
- [Derived] Serpell M, Tripathi S, Scherzinger S, Rojas-Farreras S, Oksche A, Wilson M. Assessment of Transdermal Buprenorphine Patches for the Treatment of Chronic Pain in a UK Observational Study. Patient. 2016 Feb;9(1):35-46. doi: 10.1007/s40271-015-0151-y. PMID 26547914